CLINICAL TRIAL: NCT02442700
Title: Effects of Pitavastatin on Lipid Profiles in HIV-infected Patients With Dyslipidemia and Receiving Atazanavir/Ritonavir: A Randomized, Double-blind, Crossover Study
Brief Title: Effects of Pitavastatin on Lipid Profiles in HIV-infected Patients With Dyslipidemia and Receiving Atazanavir/Ritonavir
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ramathibodi Hospital (Other)
Responsible Party: Principal Investigator, Asita Wongprikorn, Ramathibodi Hospital, Ramathibodi Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Ramathibodi Hospital 01-57-18
Record Dates: First submitted 2015-02-25; First posted 2015-05-13 (Estimated); Results first posted 2016-10-10 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-08

CONDITIONS: HIV; Dyslipidemia
Keywords: HIV-infected patients with dyslipidemia and receiving atazanavir/ritonavir
MeSH Terms: conditions — Dyslipidemias | interventions — pitavastatin

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment sequence A, B (Experimental): Treatment visits were seperated by a 2-week washout period. Treatment A = administration pitavastatin for 12 weeks; Treatment B = administration placebo for 12 weeks
  Interventions: Drug: pitavastatin; Drug: placebo
- Treatment sequence B, A (Experimental): Treatment visits were seperated by a 2-week washout period. Treatment B = adminstration placebo for 12 weeks; Treatment A = adminstration pitavastatin for 12 weeks
  Interventions: Drug: pitavastatin; Drug: placebo

INTERVENTIONS:
Drug: pitavastatin — Treatment A = administration pitavastatin for 12 weeks
  Other Names: Livalo
Drug: placebo — Treatment B = administration placebo for 12 weeks

SUMMARY:
Dyslipidemia as a risk factor for cardiovascular disease (CVD) is an increasing problem in HIV-infected patients who are on antiretroviral therapy especially protease inhibitors including atazanavir. Pitavastatin is a new HMG-CoA reductase inhibitor with lesser drug-drug interactions and demonstrable efficacy in decreasing lipid levels in non HIV-infected individuals. The study was conducted as a randomized, double-blind, crossover study comparing the safety and efficacy of pitavastatin versus placebo in HIV-infected patients with dyslipidemia and receiving atazanavir/ritonavir. Patients were randomized to receive either placebo or pitavastatin for 12 weeks, underwent a 2-week washout period, and then were given the other treatment for an additional 12 weeks. Patients were observed for lipid profiles including total cholesterol (TC), triglyceride (TG), low density lipoprotein (LDL) and high density lipoprotein (HDL); and the side effects including clinical and laboratory (serum aspartate aminotransferase (AST), alanine aminotransferase (ALT) and creatinine phosphokinase (CPK)). The follow-up visits were every 4 weeks until the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥18 years
* able to provide informed consent
* had confirmed HIV infection
* on ART including atazanavir 300 mg and ritonavir 100 mg each day in the regimens that were not changed within 12 weeks before the randomization
* patients who had cholesterol level between 200 and 500 and LDL between 130 and 400 mg/dL without any lipid-lowering agent or discontinued the lipid-lowering agent at least 1 month prior to randomization

Exclusion Criteria:

* had the history of pitavastatin and/or the constituent of the drugs allergy
* known history of myocardial infarction and/or ischemic stroke within 1 month prior to the randomization that would be endangered if we stopped the previous lipid-lowering agent before the enrollment
* abnormal AST and ALT with level ≥5 times in asymptomatic patients or ≥3 times of upper normal limit (UNL) in symptomatic patients
* pregnancy or breastfeeding
* on cyclosporine which had major drug interactions with pitavastatin
* patients who denied to join the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-05; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Asita Wongprikorn, Principal Investigator — Ramathibodi Hospital

REFERENCES:
- [Derived] Wongprikorn A, Sukasem C, Puangpetch A, Numthavej P, Thakkinstian A, Kiertiburanakul S. Effects of Pitavastatin on Lipid Profiles in HIV-Infected Patients with Dyslipidemia and Receiving Atazanavir/Ritonavir: A Randomized, Double-Blind, Crossover Study. PLoS One. 2016 Jun 15;11(6):e0157531. doi: 10.1371/journal.pone.0157531. eCollection 2016. PMID 27304841

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All subjects received all 2 treatments in a randomly assigned order. The treatments were:
  Treatment A: pitavastatin; Treatment B: placebo. The sequences were Treatments AB, BA.
Groups:
- Treatment A, B: Treatment visits were separated by a 2-week washout period. Treatment A = administration pitavastatin for 12 weeks; Treatment B = administration placebo for 12 weeks
- Treatment B, A: Treatment visits were separated by a 2-week washout period. Treatment B = administration placebo for 12 weeks; Treatment A = administration pitavastatin for 12 weeks
Period: First 12 Weeks
Arm/Group | Treatment A, B | Treatment B, A
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0
Period: Later 12 Weeks
Arm/Group | Treatment A, B | Treatment B, A
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment A, B | Treatment B, A | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.6 (10.6) | 46.7 (6.8) | 48.1 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 8 | 6 | 14
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 23.8 (2.7) | 22.5 (3.4) | 23.2 (3.1)
Underlying conditions [Number; unit: participants]
  No | 4 | 8 | 12
  Dyslipidemia | 4 | 2 | 6
  Chronic hepatitis B and C virus infection | 2 | 2 | 4
  Others | 2 | 0 | 2
Cardiovascular risk factors [Number; unit: participants]
  <2 | 7 | 11 | 18
  > or equal to 2 | 5 | 1 | 6
Baseline Creatinine [Mean (Standard Deviation); unit: mg/dL] | 0.9 (0.2) | 0.9 (0.2) | 0.9 (0.2)
Baseline Fasting blood sugar [Mean (Standard Deviation); unit: mg/dL] | 100.8 (10.1) | 97.1 (10.5) | 98.9 (10.2)
Baseline CD4 cell counts [Mean (Standard Deviation); unit: cells/mm3] | 641.9 (196.5) | 718.1 (181.2) | 680 (189)
HIV viral load <40 copies/mL [Number; unit: participants] | 12 | 11 | 23
Duration of ATV/r use [Median (Inter-Quartile Range); unit: months] | 42 [30 to 54] | 36 [24 to 36] | 36 [24 to 48]
Antiretroviral regimens combined with ATV/r [Number; unit: participants]
  TDF + FTC/3TC | 5 | 6 | 11
  TDF + other NRTIs (exclude FTC/3TC) | 2 | 2 | 4
  No TDF in backbone | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Pitavastatin in HIV-infected Patients With Dyslipidemia and Receiving Atazanavir/Ritonavir
Description: Efficacy was measured by level of TC, TG, LDL, and HDL that decreased after pitavastatin treatment. Pitavastatin was considered efficient when it could decrease TC, TG, LDL, or HDL significantly compared to placebo.
Time Frame: 12 weeks
Measure: Mean (95% Confidence Interval); unit: mg/dL
Groups:
- Treatment A: Treatment visits were separated by a 2-week washout period. Treatment A = administration pitavastatin for 12 weeks; Treatment B = administration placebo for 12 weeks
- Treatment B: Treatment visits were separated by a 2-week washout period. Treatment B = administration placebo for 12 weeks; Treatment A = administration pitavastatin for 12 weeks
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 24 | 24
mg/dL
  TC at baseline | 239.9 [220.2 to 259.6] | 257.6 [237.9 to 277.3]
  TG at baseline | 282 [123.9 to 440] | 350 [191.9 to 508]
  LDL at baseline | 144.7 [131.9 to 157.4] | 146.3 [133.6 to 159.1]
  HDL at baseline | 43 [38.1 to 47.9] | 44.8 [39.9 to 49.7]
  TC at 4 weeks after treatment | 201.3 [181.5 to 221] | 246.6 [226.9 to 266.3]
  TG at 4 weeks after treatment | 246.5 [88.4 to 404.5] | 292.5 [134.4 to 450.5]
  LDL at 4 weeks after treatment | 111.6 [98.8 to 124.4] | 142.5 [129.7 to 155.3]
  HDL at 4 weeks after treatment | 43.5 [38.6 to 48.3] | 43.5 [38.7 to 48.4]
  TC at 8 weeks after treatment | 202.3 [182.6 to 222.1] | 255.2 [235.4 to 274.9]
  TG at 8 weeks after treatment | 250.8 [92.7 to 408.8] | 334 [176 to 492.1]
  LDL at 8 weeks after treatment | 111.5 [98.7 to 124.3] | 145.1 [132.3 to 157.9]
  HDL at 8 weeks after treatment | 44.9 [40 to 49.8] | 43.7 [38.8 to 48.6]
  TC at 12 weeks after treatment | 207 [187.3 to 226.8] | 246.3 [226.5 to 266]
  TG at 12 weeks after treatment | 351.3 [193.2 to 509.4] | 279.1 [121 to 437.2]
  LDL after 12 weeks of treatment | 113.2 [100.4 to 126] | 145.6 [132.8 to 158.4]
  HDL after 12 weeks of treatment | 45.3 [40.4 to 50.2] | 44.2 [39.3 to 49.1]
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis

2. Secondary Outcome: Safety of Pitavastatin in HIV-infected Patients
Description: Safety clinical was defined by FDA; grade 1 mild symptoms; grade 2 moderate symptoms with limiting age-appropriate IADL; grade 3 severe symptoms with limiting self-care ADL, But not immediately life-threatening; grade 4 life-threatening consequences; and grade 5 death related to adverse event.
  Safety laboratory evaluation was determined safe if AST, ALT, and/or CPK level was not increased significantly comparing pitavastatin to placebo.
Time Frame: 12 weeks
Measure: Mean (95% Confidence Interval); unit: U/L
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 24 | 24
U/L
  AST at baseline | 38.2 [29.8 to 46.6] | 36.3 [27.9 to 44.7]
  ALT at baseline | 64.6 [46.7 to 82.4] | 58.9 [41 to 76.7]
  AST at 12 weeks after treatment | 39.5 [31.1 to 48] | 40.75 [32.3 to 49.2]
  ALT at 12 weeks after treatment | 64.2 [46.4 to 82.1] | 72.5 [54.6 to 90.3]

ADVERSE EVENTS:
Time Frame: 12 weeks
Groups:
- Treatment A: Treatment A = administration pitavastatin for 12 weeks
- Treatment B: Treatment B = administration placebo for 12 weeks
Arm/Group | Treatment A | Treatment B
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24

LIMITATIONS AND CAVEATS:
LImitation of this study is we did not adjust pitavastatin dosage according to lipid profiles,thus mean value of TC could not be lower than 200 mg/dL.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No